CLINICAL TRIAL: NCT07006038
Title: Vein Imaging Device on First-Attempt Success and Catheter Complications in Peripheral Intravenous Catheter Insertion
Brief Title: Vein Imaging Device on First-Attempt Success in Peripheral Intravenous Catheter Insertion
Acronym: Veinimaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Professor, Pediatric Nursing Department, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Vein Imaging-PED; 578-SBKAEK (Registry Identifier: Turkish Medicines and Medical Devices Agency)
Record Dates: First submitted 2025-05-02; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Catheterization, Peripheral; Catheters, Indwelling; Catheter Complications; Pain; Children
Keywords: pediatric emergency department; child; peripheral catheter; vein imaging device; pain; indwelling time
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The PIC insertion area was visualized with the help of the Veinlite PEDI device by the nurse. The vein imaging device was used before the PIC attempted to view the patient's veins, and after the nurse decided on the vein, the PIC was attempted.
Who Masked: Outcomes Assessor
Masking Description: The child's pain was assessed by the other non-researcher PED nurse with the FLACC pain scale.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vein imaging device group (Experimental): the PIC insertion area was visualized with the help of the device by the nurse. The vein imaging device was used before the catheter insertion attempted to view the patient's veins.
  Interventions: Device: Veinlite PEDI2
- Control group (No Intervention): no vein imaging device was used before cathater insertion

INTERVENTIONS:
Device: Veinlite PEDI2 — The Veinlite PEDI2 used before the catheter insertion.
  Arms: Vein imaging device group

SUMMARY:
This study aimed to evaluate the impact of vein visualization device on catheter placement success and catheter-related complications during peripheral IV catheter insertion in pediatric emergency departments. This randomized controlled trial compares the group using a vein visualization device with the group using the standard method.

DETAILED DESCRIPTION:
There were two groups in this study: the vein imaging device and the control group.

The children to be included in this study consisted of pediatric patients who were admitted to the PED. There were two groups in this study: the vein imaging device and the control group. If the physician requested a peripheral intravenous catheter (PIC), the vein imaging device was applied to increase the first-attempt success of the PIC in one group. In addition, there was a control group in which any device was not used. One trained nurse who was a PhD student enrolled the participants who met the eligibility criteria.

The patients who were scheduled for PIC insertion were allocated to groups according to the randomization scheme. After providing information to the child and the parent, the investigator obtained consent from the parent, and the group assignment was determined. The patients in the control group did not receive any additional interventions and were observed during the PIC insertion after obtaining consent.

The PIC procedure time started when the tourniquet connected. In the vein imaging device and the control groups, communication with the child was maintained using the questions mentioned above during the procedure by the researcher nurse. When the phlebotomist nurse decided on the insertion site for the PIC, the PIC was attempted. If the PIC was inserted on the first attempt, the PIC procedure time stopped. If not, when the PIC was successfully inserted, the PIC procedure time was stopped. The PIC insertion time was recorded in minutes for successful PIC insertion. After the PIC insertion area was closed with dressing and the materials were collected, the child's pain was assessed by the PED nurse with the FLACC pain scale.

Complication signs and symptoms are monitored in the PIC area. If the PIC is to be removed for any reason, the reason and time of removal are recorded. PIC indwelling time was recorded. If it was removed due to a complication, the PIC area was followed up by grading with infiltration, extravasation, and phlebitis scales.

ELIGIBILITY:
Inclusion Criteria:

* The physician must inform them that PIC must be inserted to administer medication and fluids
* The parent must voluntarily agree to participate in the study, consent form must be obtained from the parent

Exclusion Criteria:

* The child presenting to the pediatric emergency department must be in shock or severely dehydrated, requiring urgent intervention
* No need for PIC
* Presence of a central venous catheter (since there will be no need for PIC)
* Selection of the lower extremities for PIC placement (since they may experience more pain and complication)
* Use of sedatives or analgesics before the PIC procedure (at least 4 hours before)

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 206 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
PIC insertion success | through the PIC insertion
  first-attempt PIC insertion success
procedural time | through the PIC insertion
  procedural time for successful PIC insertion

SECONDARY OUTCOMES:
PIC insertion related pain score | FLACC score evaluated 3 minutes after the PIC insertion
  The FLACC (Face, Legs, Activity, Cry, Consolability) score related to the PIC insertion. The scale is scored in a range of 0-10, with 0 representing no pain. Assessment of score:
  0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
PIC indwelling time | through the PIC stay (If the PIC is to be removed for any reason, the reason and time of removal are recorded, PIC indwelling time was recorded as hours)
  PIC stay time

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, Assoc. Prof., Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)